CLINICAL TRIAL: NCT03769246
Title: Upright Back Posture Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Upright Technologies (Industry)
Responsible Party: Principal Investigator, Joel Stein, MD, Professor of Physical Medicine and Rehabilitation; Chair of Department of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAR4123
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Back Pain; Postural Low Back Pain; Lower Back Pain
Keywords: Upright; Back; Posture; Back pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Upright Go Device Group (Experimental): Patients receiving the Upright device will have a brief training on the use of the device and proper posture. They will be asked to download the Upright app on their phone from the Playstore.
  Patients will wear the device once daily for training. They will attach the device applying an adhesive on their upper back, as instructed, and the device will be attached to the adhesive by velcro. Once completed they should remove adhesive.
  Interventions: Device: Upright Go Device
- Control Group (Active Comparator): The control group will receive a 15-20 minute instruction on proper posture by the physician and will receive an ergonomic handout.
  Interventions: Other: Ergonomic Handout

INTERVENTIONS:
Device: Upright Go Device — Participants will be asked to use the Upright device everyday for four (4) weeks. After four (4) weeks, the participants will be asked to complete a couple of questionnaires regarding their pain scale and back posture.
  Other Names: Upright Technologies
  Arms: Upright Go Device Group
Other: Ergonomic Handout — Participants will be asked to use the ergonomic handout everyday for four (4) weeks. After four (4) weeks, the participants will be asked to complete a couple of questionnaires regarding their pain scale and back posture.
  Arms: Control Group

SUMMARY:
This is a randomized controlled study to determine if patients between the ages of 18-50 years, with posture related low back pain, who use the Upright device demonstrate improved pain control and self perception of posture compared to those given standard ergonomic instruction.

DETAILED DESCRIPTION:
Back pain is a common complaint among students. For many, back pain is directly related to poor posture while sitting and standing. Those who spend prolonged time sitting in poor posture often develop muscular imbalances leading to tight chest muscles and weakness in back muscles. The Upright system is a device which helps provide a sensory reminder to alert users when their posture is poor. The purpose of this study is to determine if patients who use the upright posture device demonstrate improved pain control and self perception of posture when compared to those given standard ergonomic instruction.

ELIGIBILITY:
Inclusion Criteria:

* Postural-related back pain

Exclusion Criteria:

* A diagnosis of significant scoliosis, herniated/bulging disc, lumbar spondylolysis, radiculitis, facet arthrosis, fibromyalgia, rheumatoid arthritis, seronegative spondyloarthropathy.
* Neurologic deficits on exam
* Currently in physical therapy (PT)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Christina Bevelaqua, M.D, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Upright Go Device Group: Patients receiving the Upright device will have a brief training on the use of the device and proper posture. They will be asked to download the Upright app on their phone from the Playstore.
  Patients will wear the device once daily for training. They will attach the device applying an adhesive on their upper back, as instructed, and the device will be attached to the adhesive by velcro. Once completed they should remove adhesive.
  Upright Go Device: Participants will be asked to use the Upright device everyday for four (4) weeks. After four (4) weeks, the participants will be asked to complete a couple of questionnaires regarding their pain scale and back posture.
Period: Overall Study
Arm/Group | Upright Go Device Group | Control Group
Started | 15 | 15
Completed | 13 | 15
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upright Go Device Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (6.6) | 30.2 (7.1) | 29.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Postural Back Pain [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Score on Numeric Pain Rating Scale (NPRS)
Description: The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). Averages were taken of each group, pre and post intervention. A higher score represents a worse outcome, and a lower score represents a better outcome.
Time Frame: 4 weeks
Population: Two subjects in the Upright Go Device Group were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upright Go Device Group | Control Group
Number analyzed (Participants) | 15 | 15
score on a scale
  NPRS Pre | 2.54 (1.81) | 2.44 (1.99)
  NPRS Post: number analyzed (Participants) | 13 | 15
  NPRS Post | 1.75 (1.45) | 1.49 (1.17)

2. Primary Outcome: Score on the PROMIS Pain Interference Short Form 6b
Description: The Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference Short Form utilizes a 7-day recall period (items include the phrase "In the past 7 days..."). Individuals are to score pain interference for each of the 6 questions from a scale of 1 to 5.
  1. = Not at all
  2. = A little bit
  3. = Somewhat
  4. = Quite a bit
  5. = Very Much
  Scores are collected and analyzed as individual questions, and not as an aggregate total. Averages were taken of each question, for each group, pre and post intervention. A higher score represents a worse outcome and a lower score represents a better outcome.
Time Frame: 4 weeks
Population: Two subjects in the Upright Go Device Group were lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upright Go Device Group | Control Group
Number analyzed (Participants) | 15 | 15
score on a scale
  Responses to Question 1: "How much did pain interfere with your enjoyment of life?" (Pre) | 2.40 (1.06) | 2.53 (1.19)
  Responses to Question 1: "How much did pain interfere with your enjoyment of life?" (Post): number analyzed (Participants) | 13 | 15
  Responses to Question 1: "How much did pain interfere with your enjoyment of life?" (Post) | 1.85 (0.90) | 1.60 (0.51)
  Responses to Question 2: "How much did pain interfere with your ability to concentrate?" (Pre) | 2.27 (1.03) | 2.47 (1.06)
  Responses to Question 2: "How much did pain interfere with your ability to concentrate?" (Post): number analyzed (Participants) | 13 | 15
  Responses to Question 2: "How much did pain interfere with your ability to concentrate?" (Post) | 1.69 (0.63) | 1.67 (0.62)
  Responses to Question 3: "How much did pain interfere with your day to day activities?" (Pre) | 2.40 (1.24) | 2.53 (1.19)
  Responses to Question 3: "How much did pain interfere with your day to day activities?" (Post): number analyzed (Participants) | 13 | 15
  Responses to Question 3: "How much did pain interfere with your day to day activities?" (Post) | 1.62 (0.96) | 1.67 (0.62)
  Responses to Q4: "How much did pain interfere with your enjoyment of recreational activities?" (Pre) | 2.33 (1.11) | 2.47 (1.06)
  Responses to Q4:"How much did pain interfere with your enjoyment of recreational activities?" (Post): number analyzed (Participants) | 13 | 15
  Responses to Q4:"How much did pain interfere with your enjoyment of recreational activities?" (Post) | 1.54 (0.78) | 1.40 (0.51)
  Responses to Question 5: "How much did pain interfere with doing your tasks away from home?" (Pre) | 2.20 (0.86) | 2.40 (1.35)
  Responses to Question 5:"How much did pain interfere with doing your tasks away from home?" (Post): number analyzed (Participants) | 13 | 15
  Responses to Question 5:"How much did pain interfere with doing your tasks away from home?" (Post) | 1.69 (0.63) | 1.33 (0.62)
  Responses to Question 6: "How often did pain keep you from socializing with others?" (Pre) | 1.73 (0.88) | 1.47 (0.83)
  Responses to Question 6: "How often did pain keep you from socializing with others?" (Post): number analyzed (Participants) | 13 | 15
  Responses to Question 6: "How often did pain keep you from socializing with others?" (Post) | 1.15 (0.38) | 1.13 (0.35)

ADVERSE EVENTS:
Time Frame: Participants participated in the study for a total of 4 weeks, or 1 month.
Arm/Group | Upright Go Device Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT03769246/Prot_SAP_002.pdf